CLINICAL TRIAL: NCT06153563
Title: Evaluation of the Elasticity of the Mitral Valve Chordae by Uniaxial Traction in the Context of Mitral Valve Regurgitation With a Comparison of the Results: Mitral Valve Prolapse vs Restriction of Mitral Valve Movement
Brief Title: Evaluation of the Elasticity of the Mitral Valve
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN1102022/CHUSTE
Record Dates: First submitted 2023-11-23; First posted 2023-12-01 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Mitral Valve Disease
Keywords: Mitral valve; mitral valve chords; elasticity; Young's modulus; mitral valve histology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mitral valve prolapse: Patients with mitral valve prolapse
  Interventions: Other: Data collection on patient history and intraoperative results.
- Restrictive ischemic mitral valve: Patients with restrictive ischemic mitral valve
  Interventions: Other: Data collection on patient history and intraoperative results.

INTERVENTIONS:
Other: Data collection on patient history and intraoperative results. — Data collection on patient history and intraoperative results.

SUMMARY:
There is no information in the literature on the mechanobiological characteristics of mitral valve chords in living humans. All examinations were carried out on tissues taken from animals, either from cadavers or from frozen human tissues. The objective is to determine mechanobiological and histological characteristics of the mitral valve chords in living humans, as well as to compare differences in elasticity in different groups (Group A: patients with mitral valve prolapse versus Group B: patients with restrictive ischemic mitral valve).

DETAILED DESCRIPTION:
The prospective study will be conducted on 20 patients, who will be selected consecutively without randomization. The inclusion and exclusion criteria are determined.

The harvested tissue will not be frozen and will kept in natural conditions as close as possible.

ELIGIBILITY:
Inclusion Criteria:

All patients programmed for mitral valve replacement who have more than 45 years old

Exclusion Criteria:

* Patients with mitral calcification
* Mitral valve rheumatic disease
* Mitral valve infections
* Redo surgery on the mitral valve

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients programmed for mitral valve replacement who have more than 45 years old
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Maximum value of Young's modulus | Hour 1
  Comparison of elasticity difference between the two groups

SECONDARY OUTCOMES:
First histological evaluation | Hour 1
  Determine the histological characteristics of living humans

CONTACTS AND LOCATIONS:
Overall Officials: Andranik PETROSYAN, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No